CLINICAL TRIAL: NCT02096900
Title: A Comparison of Midazolam and Zolpidem as Oral Premedication in Children
Acronym: PedsPreMed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Davinder Ramsingh, MD, Principal Investigator, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5140032
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Parental/Caregiver Anxiety; Child's Anxiety
Keywords: Pre-medication; Pre-operative anxiety
MeSH Terms: interventions — Zolpidem; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zolpidem (Active Comparator): zolpidem given orally 0.25mg/kg pre-operatively single dose
  Interventions: Drug: zolpidem
- midazolam (Active Comparator): midazolam will be given at 0.5mg/kg, pre-operatively single dose
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: zolpidem — Zolpidem will be given one time at 0.25 mg/kg pre-operatively
  Other Names: ambien
  Arms: zolpidem
Drug: Midazolam
  Other Names: versed
  Arms: midazolam

SUMMARY:
The purpose of this investigator-initiated study is to compare the efficacy of oral midazolam and zolpidem for preoperative sedation, anxiety of patient, and caregiver anxiety at the time of separation, and ease of mask acceptance at induction in children. Subjects will be randomized to receive oral medication midazolam or zolpidem approximately 30 minutes prior to surgery. No placebo will be administered in this study. Subjects will be male and female children between 2 and 9 years of age. In total, subject participation will last approximately the duration of their preoperative, perioperative, and immediate postoperative period. A member of the research team will recruit subjects preoperatively in the operating room holding area prior to surgery. Consent will take place at the time of recruitment in the preoperative holding area following a detailed explanation of the study and medications involved in the study. Participants will be of ASA (American Society of Anesthesiologists) class I-II, undergoing surgical procedures of at least 2 hours duration, and expected to remain inpatient for at least 23 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ages 2-9 years
* ASA class I-II
* inpatient surgeries of at least 2 hours duration
* requiring postoperative admission of at least 23 hours Exclusion Criteria:

Exclusion Criteria:

* contraindication to preoperative sedation, known allergy or sensitivity to the study medications,
* those who lack legal representative consent
* Patients with weights lying below the 5th percentile or above the 95th percentile according to the current published CDC growth chart will also be excluded regardless of existing specific contraindication.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2016-05-06 (Actual); Study Completion 2016-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amgad Hanna, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Midazolam: midazolam was given at 0.5mg/kg, pre-operatively single dose
- Zolpidem: zolpidem was given orally 0.25mg/kg pre-operatively single dose
Period: Overall Study
Arm/Group | Midazolam | Zolpidem
Started | 42 (Allocated to Midazolam) | 44 (Allocated to Zolpidem)
Completed | 38 | 42
Not Completed | 4 | 2
Not completed — Did not receive medication | 3 | 1
Not completed — Surgery cancelled- medication received | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analyses subjects who completed the study per protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Zolpidem | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.34 (2.21) | 6.07 (2.34) | 6.20 (2.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 17 | 23 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 25 | 47
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 2 | 2
  White | 36 | 40 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 42 | 80
Weight (kg) [Mean (Standard Deviation); unit: kg] | 23.16 (6.20) | 23.18 (7.21) | 23.17 (6.71)
Height (cm) [Mean (Standard Deviation); unit: cm] | 117.32 (14.55) | 115.34 (15.92) | 116.29 (15.23)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 16.73 (1.92) | 17.60 (4.02) | 17.19 (3.21)
ASA physical status [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) physical status classification system provides assessment of the fitness of patients before surgery.
  ASA PS I patient is a normal healthy patient. ASA PS II patient is a patient with mild systemic disease without substantive functional limitations, for example; well controlled diabetes/hypertension or mid lung disease.
  Participants
    ASA PS I | 12 | 14 | 26
    AS PS II | 26 | 28 | 54
Time from drug administration to parental separation (minutes) [Mean (Standard Deviation); unit: minutes] | 31.53 (12.20) | 34.98 (16.00) | 33.13 (14.31)
Duration of anesthesia (minutes) [Mean (Standard Deviation); unit: minutes] | 185.58 (72.20) | 205.79 (97.60) | 196.46 (86.86)

OUTCOME MEASURES:

1. Primary Outcome: Patient Anxiety at the Time of Separation
Description: The primary outcome measure of patient anxiety will be measured using the validated Modified Yale Preoperative Anxiety Score (mYPAS). The mYPAS is the current standard for evaluation of anxiety in children receiving anesthesia for surgical procedures.
  The modified Yale Preoperative Anxiety scale (m-YPAS) is a structured observational measure of preoperative anxiety in children. It was developed by the study group lead by Kain Z. It consists of assessment of 27 items in 5 domains of behavior indicating anxiety in young children; activity, emotional expressivity, state of arousal, vocalization, and use of parents. Each item is weighted in calculation of the total score that ranges from 22.5 -100. Children with a score above 30 are considered anxious while those with the score of 30 or less were considered not anxious.
Time Frame: Up to 24 hours including preoperative, preoperative, and postoperative periods.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Midazolam | Zolpidem
Number analyzed (Participants) | 38 | 42
units on a scale | 26.69 [23.30 to 36.60] | 30.00 [23.30 to 38.20]

2. Secondary Outcome: Mask Acceptance Score
Description: Mask acceptance by the patient, will be measured on a 4-point scale adapted from a similar trial.
  Score of 1 and 2 indicates satisfactory mask acceptance. Score of 3 or 4 indicates unsatisfactory mask acceptance during induction of general anesthesia.
Time Frame: During induction of general anesthesia.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Zolpidem
Number analyzed (Participants) | 38 | 42
Participants
  Mask acceptance score 1-2 | 34 | 29
  Mask acceptance score 3-4 | 4 | 13

3. Secondary Outcome: Presence of Emergence Delirium During Recovery
Description: Presence or absence of emergence delirium during recovery, will be assessed using the pediatric anesthesia emergence delirium (PAED) scale recorded at 5-minute intervals for 20 minutes following the child's spontaneous eye opening. PAED score of ≥12 at any time indicates presence of emergence delirium.
Time Frame: Up to 30 minutes after child's first eye opening in the post-operative period.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Zolpidem
Number analyzed (Participants) | 38 | 42
Participants
  No | 26 | 32
  Yes | 12 | 10

4. Secondary Outcome: Parental/Caregiver Anxiety Assessed Using the Validated State-Trait Anxiety Inventory for Adults (STAI)
Description: Parental/caregiver anxiety, was assessed using the validated State-Trait Anxiety Inventory for Adults (STAI), a validated self-evaluation questionnaire.
  The STAI is compromised of separate self-report scales for measuring state and trait anxiety. The S-Anxiety scale (STAI Form Y-1) consists of twenty statements that evaluate how respondents feel "right now, at this moment". The T-Anxiety scale (STAI Form Y-2) consists of twenty statements that assess how respondents generally feel. The score ranges from 20 (most relaxed) to 80 (highest stress).
  The baseline STAI inventory was completed by e parent/caregiver after obtaining the informed consent in the preoperative holding area and before the subject was separated from the caregiver. Baseline STAI inventory consisted of form STAIY-1 (State Anxiety) and form STAIY-2 (Trait Anxiety) anxiety.
  After caregiver/patient separation,form STAIY-1(State Anxiety) was completed again by the caregiver.
Time Frame: Preoperative holding area from the time of informed consent until caregiver/patient separation.
Population: only total of 51 subjects were analyzed. Caregivers of 29 subjects were given incorrect form to fill at time of separation rendering data not applicable for analysis for the 29 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midazolam | Zolpidem
Number analyzed (Participants) | 24 | 27
units on a scale
  STAIY-1 (at informed consent) | 41.74 (10.66) | 41.12 (10.88)
  STAIY-2 (at informed consent) | 31.81 (8.29) | 34.12 (8.29)
  STAIY-1 (at separation) | 44.33 (9.58) | 43.85 (13.70)

5. Post Hoc Outcome: Modified Yale Preoperative Anxiety Scale (mYPAS) Score at Separation (mYPAS2) Based on Baseline (mYPAS1) Score.
Description: Midazolam group participants will be separated into two groups; non-anxious (mYPAS1 ≤ 30) at baseline and anxious (mYPAS1 > 30) at baseline. The mYAPS2 scores of these two groups will be compared to the mYPAS2 scores of the Zolpidem group participants.
  The modified Yale Preoperative Anxiety scale (m-YPAS) is a structured observational measure of preoperative anxiety in children that takes less than a minute to preform. It consists of assessment of 27 items in 5 domains of behavior indicating anxiety in young children; activity, emotional expressivity, state of arousal, vocalization, and use of parents. Each item is weighted in calculation of the total score that ranges from 22.5 -100. A cut off 30 on the m-YPAS scale was found to balance the high specificity and sensitivity while maintaining high positive predictive value. Children with a score above 30 are considered anxious while those with the score of 30 or less were considered not anxious.
Time Frame: Up to 24 hours including pre-operative, peri-operative and post-operative periods.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Midazolam | Zolpidem
Number analyzed (Participants) | 38 | 42
units on a scale
  mYPAS2 - non-anxious baseline | 23.32 [23.30 to 30.80] | 28.30 [23.30 to 42.50]
  mYPAS2 - anxious baseline | 29.97 [23.30 to 46.60] | 60.75 [36.60 to 96.70]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the study participation time which was about one day for each subject.
Arm/Group | Midazolam | Zolpidem
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/42
Other Adverse Events (participants affected / at risk) | 1/38 | 5/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=38) | Zolpidem (N=42)
Oxygen desatruation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Oxygen desaturation with pulse oximeter reading less than 94% for 33 seconds (SPO2 range 87-94%). Resolved when deep breathing was encouraged.
Double vision (Nervous system disorders) | 0 (0) | 2 (2)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Epigastric pain. Likely related to preoperative fasting rather than the investigational drug.
Visual Hallucinations (Nervous system disorders) | 0 (0) | 2 (2)
Involuntary tongue movements (Nervous system disorders) | 0 (0) | 1 (1)
Dysphoria (Nervous system disorders) | 0 (0) | 1 (1) — Unpleasant sensation after taking the medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes